CLINICAL TRIAL: NCT00970008
Title: Exploring Massage Benefits for Arthritis of the Knee
Acronym: EMBARK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AT004623-01 (NIH)
Record Dates: First submitted 2009-08-18; First posted 2009-09-02 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Massage 30 min - 2x wk for 4 wks & 1x wk for 4 wks (Active Comparator): Swedish massage session of 30 minutes duration, twice weekly for four weeks followed by once weekly for four weeks over a eight (8) week period. Total intervention = 12 sessions for 360 minutes.
  Interventions: Other: Massage 30 min 2x/wk x4 wks then 1x/wk x4 wks
- Massage 60 min - 2x wk for 4 wks & 1x wkly for 4 wks (Active Comparator): Swedish massage session of 60 minutes duration, twice weekly for four weeks followed by once weekly for four weeks over a eight (8) week period. Total intervention = 12 sessions for 720 minutes.
  Interventions: Other: Massage 60 min 2x/wk for 4 wks then 1x/wk for 4 wks
- Massage 30 min sessions - 1x/wk for 8wks (Active Comparator): Swedish massage session of 30 minutes duration, once weekly for eight weeks over a eight (8) week period. Total intervention = 8 sessions for 240 minutes.
  Interventions: Other: Massage 30 min sessions 1x/wk for 8 wks
- Massage 60 min sessions - 1x/wk for 8 wks (Active Comparator): Swedish massage session of 60 minutes duration, once weekly for eight weeks over a eight (8) week period. Total intervention = 8 sessions for 480 minutes
  Interventions: Other: Massage 60 min session 1x/wk for 8 wks
- Usual Care Control (No Intervention): Continue on usual care for eight (8) week period.

INTERVENTIONS:
Other: Massage 30 min 2x/wk x4 wks then 1x/wk x4 wks — Swedish massage session of 30 minutes duration, twice weekly for four weeks followed by once weekly for four weeks over a eight (8) week period. Total intervention = 12 sessions for 360 minutes.
  Arms: Massage 30 min - 2x wk for 4 wks & 1x wk for 4 wks
Other: Massage 60 min 2x/wk for 4 wks then 1x/wk for 4 wks — Swedish massage session of 60 minutes duration, twice weekly for four weeks followed by once weekly for four weeks over a eight (8) week period. Total intervention = 12 sessions for 720 minutes.
  Arms: Massage 60 min - 2x wk for 4 wks & 1x wkly for 4 wks
Other: Massage 30 min sessions 1x/wk for 8 wks — Swedish massage session of 30 minutes duration, once weekly for eight weeks over a eight (8) week period. Total intervention = 8 sessions for 240 minutes.
  Arms: Massage 30 min sessions - 1x/wk for 8wks
Other: Massage 60 min session 1x/wk for 8 wks — Swedish massage session of 60 minutes duration, once weekly for eight weeks over a eight (8) week period. Total intervention = 8 sessions for 480 minutes
  Arms: Massage 60 min sessions - 1x/wk for 8 wks

SUMMARY:
In 2004, we conducted a pilot randomized, wait list controlled, trial (RCT) of massage therapy for OA of the knee in 68 subjects. That study, supported by CDC grant SIP-14-00, revealed the potential efficacy of Swedish massage therapy in the treatment of OA of the knee, with benefits of increased function and decreased pain persisting at least eight weeks following treatment cessation. The results of that trial, the first RCT of massage for OA, were published in the Archives of Internal Medicine in 2006 (See reference in More Information section). This current project builds on the design and findings of the pilot trial to determine the optimal dose and treatment regimen and provide longer term follow up. This project is a dual-site, randomized, dose-ranging trial to compare four dose/regimens in order to identify the optimal protocol for clinical practice.

The primary study hypothesis is that an eight (8) week course of Swedish massage therapy of one of the four proposed doses (by frequency and duration of massage treatment session) will be effective in reducing pain and improving function in patients with confirmed OA of the knee.

DETAILED DESCRIPTION:
A dual-site, randomized, dose-ranging trial to determine the role and practice parameters for massage in the standard clinical management of OA based on investigation of efficacy and mechanism of action. The study hypothesis is that an 8 week course of Swedish massage therapy will be effective in reducing pain and improving function in patients with confirmed OA of the knee. A future phase III trial is planned to test the optimal massage intervention identified in this study against a validated sham/control intervention, incorporating all pertinent outcome measures from the antecedent studies. In addition, this study will further the development of robust methodologies to test the efficacy of massage interventions in general. The research agenda advanced by the current study will culminate with the establishment of the proper place for massage therapy among standard treatment options for the millions of Americans suffering with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* 35 years of age or greater.
* Written confirmation of OA of the knee as provided by the participant's physician.
* Radiographically-established OA of the knee.
* Pre-randomization score of 40 to 90 on the Visual Analog Pain Scale (0-100 mm scale).
* Patients with bilateral knee involvement will have the more severely affected knee designated as the study knee.
* American College of Rheumatology defined OA of the knee:

  1. Knee pain
  2. Satisfaction of at least five of the following nine criteria:

  <!-- -->

  1. Age greater than 50 years
  2. Stiffness < 30 minutes
  3. Crepitus
  4. Bony tenderness
  5. Bony enlargement
  6. No palpable warmth
  7. ESR < 40 mm/hr
  8. Rheumatoid Factor (RF) < 1:40

Exclusion Criteria: (no exclusion criterion may be present)

* Presence of rheumatoid arthritis, fibromyalgia, recurrent or active pseudo gout.
* Presence of cancer or other serious medical conditions.
* Signs or history of kidney or liver failure.
* Presence of asthma requiring the use of corticosteroid treatment.
* Use of oral corticosteroids within the past four weeks.
* Use of intra-articular knee depo-corticosteroids with the past three months.
* Use of intra-articular hyaluronate with the past six months.
* Arthroscopic surgery of the knee within the past year.
* Significant injury to the knee within the past six months.
* Presence of a rash or open wound over the knee.
* Unable to satisfy the treatment and follow-up requirements.
* Unable to provide written informed consent.
* Currently receiving massage therapy on a regular basis (at least twice a month).
* Knee replacement of study knee (ok if the knee not being studied has been replaced).

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Improvement in WOMAC (Western Ontario Multipurpose Arthritis Centers) Knee and Hip Osteoarthritis Index | Six (6) months

SECONDARY OUTCOMES:
Safety | Six (6) months
Improvement in range of motion as measured by a goniometer. | six (6) months
Improvement in physical function as measured by time in seconds to walk fifty (50) feet on a level straight surface. | six (6) months
Reduction in pain as measured by the Visual Analog Scale (VAS) for pain. | Six (6) months

CONTACTS AND LOCATIONS:
Overall Officials: Adam I Perlman, MD, MPH, Principal Investigator — University of Medicine and Dentistry of New Jersey
Locations (2):
- United States (2):
  - Yale-Griffin Prevention Research Center/Griffin Hospital, Derby, Connecticut
  - Siegler Center for Integrative Medicine - Saint Barnabas Ambulatory Care Center, Livingston, New Jersey

REFERENCES:
- [Background] Perlman AI, Sabina A, Williams AL, Njike VY, Katz DL. Massage therapy for osteoarthritis of the knee: a randomized controlled trial. Arch Intern Med. 2006 Dec 11-25;166(22):2533-8. doi: 10.1001/archinte.166.22.2533. PMID 17159021
- [Derived] Ali A, Kahn J, Rosenberger L, Perlman AI. Development of a manualized protocol of massage therapy for clinical trials in osteoarthritis. Trials. 2012 Oct 4;13:185. doi: 10.1186/1745-6215-13-185. PMID 23035641
- [Derived] Perlman AI, Ali A, Njike VY, Hom D, Davidi A, Gould-Fogerite S, Milak C, Katz DL. Massage therapy for osteoarthritis of the knee: a randomized dose-finding trial. PLoS One. 2012;7(2):e30248. doi: 10.1371/journal.pone.0030248. Epub 2012 Feb 8. PMID 22347369